CLINICAL TRIAL: NCT04287374
Title: The Effects of Online Single-Session Interventions on College Student Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 834854
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Well-Being; Depressive Symptoms; Anxiety; Affect
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component Well-being Intervention (Experimental): Reading and writing activities based on cognitive restructuring (rephrasing automatic negative thoughts), gratitude (noticing and appreciating good things in life), and behavioral activation (identifying and scheduling positive activities)
  Interventions: Behavioral: Multi-component Well-being Intervention
- Study Skills Control (Sham Comparator): Reading and writing activities designed to teach evidence-based study strategies.
  Interventions: Behavioral: Study Skills

INTERVENTIONS:
Behavioral: Multi-component Well-being Intervention — The intervention asks participants to complete exercises based on three different skills. These skills include cognitive restructuring, gratitude and behavioral activation. After completing the program, participants will pick their favorite exercise to complete on a weekly basis for homework. In order to increase compliance with the homework, participants will complete a short plan in which they will identify when, where and with who they will complete the homework. The whole intervention takes approximately 20-30 minutes to complete.
  Arms: Multi-component Well-being Intervention
Behavioral: Study Skills — Participants are taught three different study skills/strategies. They are asked to make a plan to continue using these strategies after completing the intervention. The whole intervention takes approximately 20-30 minutes to complete.
  Arms: Study Skills Control

SUMMARY:
This study seeks to investigate the effects of an online single-session intervention on college student mental health and well-being. Undergraduate students from the University of Pennsylvania and Harvard will be randomized to a 30-minute single-session intervention or a study skills control group. Students' depressive symptoms, anxiety symptoms, positive and negative affect, and subjective well-being will be assessed up to 12 weeks post-intervention.

DETAILED DESCRIPTION:
The design of our study is a randomized control trial. After enrollment in the study, participants will randomly assigned to one of two conditions. In each condition, participants will be asked to complete an initial survey of mental health and well-being measures. Following this survey, participants will complete either a well-being skills single-session intervention or control single-session intervention (study skills) depending on which condition they were assigned to. These single-session interventions educate the participant on their focal concept and teach them exercises to improve that skill. Completing the single-session intervention will take approximately 20-30 minutes.

After completing their single-session intervention, all participants will retake the measures of mental health and well-being presented to them at the beginning of the program. Participants will also be asked to complete measures of intervention feasibility, acceptability and appropriateness at this time.

Following this initial intervention, participants will retake the measures of well-being and mental health at 2 weeks, 4 weeks, and 12 weeks after they completed the intervention. This will allow us to fulfill our first objective by determining how long single-session interventions improve undergraduate mental health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Current undergraduate student at select universities
* Able to access the internet
* Can participate in follow-up surveys for three months post sign-up

Exclusion Criteria:

* Unable to access the internet
* Will not be able to respond to the follow-up surveys post-intervention

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Depression Questionnaire. The total score ranges from 0 to 27. Lower scores indicate a better outcome.
Change in Generalized Anxiety Disorder Screener-7 (GAD-7) | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
Change in The Warwick-Edinburgh Mental Wellbeing Scale | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Well-being questionnaire. Total score ranges from 14 to 70. Higher values indicate a better outcome.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | Immediately post-intervention (0 weeks)
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Feasibility of Intervention Measure | Immediately post-intervention (0 weeks)
  Questionnaire measuring the feasibility of an intervention. Feasibility refers to the degree to which a treatment can be successfully implemented in a given setting. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Intervention Appropriateness Measure | Immediately post-intervention (0 weeks)
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Change in Gratitude Questionnaire-6 | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Gratitude questionnaire. Total score ranges from 6 to 42. Higher scores indicate more gratitude.
Change in Beck Hopelessness Scale (4-item version) | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Hope Questionnaire. Total score ranges from 0 to 4. Higher scores indicate less hope (or more hopelessness).
Change in Perceived Stress Scale-4 | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Perceived stress questionnaire. Total score ranges from 0 to 16. Higher scores indicate more stress.
Change in Positive and Negative Affect Schedule | Change from baseline at 2 week follow-up, 4 week follow-up, 12 week follow-up
  Affect Questionnaire. Scores range from 10-50 for positive affect and negative affect subscales. Higher scores represent higher levels of affect.

CONTACTS AND LOCATIONS:
Overall Officials: Robert DeRubeis, PhD, Study Director — University of Pennsylvania; Akash Wasil, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Harvard University, Cambridge, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No